CLINICAL TRIAL: NCT07085000
Title: Preoperative Cognitive and Physical Frailty as Predictors of Decision Satisfaction and Postoperative Adaptation in Geriatric Gynecologic Oncology Patients: A Pilot Observational Study
Brief Title: Cognitive and Physical Frailty as Predictors of Decision Satisfaction in Geriatric Gynecologic Oncology
Acronym: GYNCOGFRAIL
Status: Completed | Type: Observational
Sponsor: Izmir City Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: ISHGGO
Record Dates: First submitted 2025-07-16; First posted 2025-07-25 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Gynecologic Cancer; Frailty; Cognitive Impairment; Geriatric Oncology
Keywords: Cognitive Function; Frailty; MoCA; CFS; Decision Satisfaction; Postoperative Recovery; Geriatric Patients; Gynecologic Surgery; Patient-Reported Outcomes
MeSH Terms: conditions — Frailty; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Geriatric Gynecologic Cancer Patients: This cohort includes female patients aged 65 years or older with a diagnosis of gynecologic malignancy who are scheduled for elective surgery. Cognitive status and physical frailty will be assessed preoperatively, and participants will be followed postoperatively to evaluate decision satisfaction and adaptation parameters.
  Interventions: Other: No Intervention - Observational Assessment

INTERVENTIONS:
Other: No Intervention - Observational Assessment — No intervention is applied. Preoperative cognitive status (MoCA) and physical frailty (CFS) are assessed as part of observational data collection. Postoperative follow-up includes decision satisfaction and adherence evaluations.

SUMMARY:
This prospective observational study aims to evaluate the association between preoperative cognitive function, measured by the Montreal Cognitive Assessment (MoCA), and physical frailty, assessed using the Clinical Frailty Scale (CFS), with postoperative decision satisfaction and adaptation in geriatric patients undergoing gynecologic cancer surgery. Approximately 60 to 70 female patients aged 65 years or older will be enrolled. Participants will complete preoperative assessments of cognitive status and frailty. Postoperative outcomes including decision satisfaction, medication adherence, mobilization, respiratory exercise compliance, and return to functional baseline will be evaluated. The study is conducted at İzmir City Hospital and is designed to generate preliminary data to inform larger-scale research.

DETAILED DESCRIPTION:
The study is designed as a prospective observational investigation involving geriatric female patients diagnosed with gynecologic cancers, including endometrial, ovarian, cervical, and vulvar malignancies. All participants are scheduled for elective surgical procedures at İzmir City Hospital. The primary objective is to explore the relationship between preoperative cognitive status, assessed by the Montreal Cognitive Assessment (MoCA), and physical frailty, assessed by the Clinical Frailty Scale (CFS), with postoperative decision satisfaction and multidimensional adaptation.

Decision satisfaction will be measured using the Decision Regret Scale (DRS) within the first postoperative week. Postoperative adaptation will be evaluated through a composite score that includes early mobilization, adherence to respiratory exercises (such as incentive spirometry), medication adherence, attendance at follow-up appointments, and return to baseline functional capacity, assessed at postoperative day 30.

Approximately 60 to 70 participants will be enrolled. Data will be analyzed using descriptive statistics, correlation analysis, and multivariable regression to identify the predictive value of cognitive and frailty assessments on postoperative outcomes. The findings are expected to contribute to the development of personalized perioperative care strategies for older adults with gynecologic cancers.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 65 years or older
* Diagnosed with a gynecologic malignancy (endometrial, ovarian, cervical, or vulvar cancer)
* Scheduled for elective surgery with curative or staging intent
* Ability to provide informed consent
* Ability to complete preoperative cognitive (MoCA) and frailty (CFS) assessments

Exclusion Criteria:

* Diagnosis of severe dementia or MoCA score <10
* Undergoing emergency surgery
* Patients under exclusive palliative care
* Non-Turkish speaking or inability to comprehend study assessments
* Presence of severe psychiatric conditions interfering with cognitive assessment

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes — Only biologically female patients are eligible to participate, regardless of gender identity.
Study Population: Older female patients diagnosed with gynecologic malignancies who are scheduled for elective surgery at İzmir City Hospital. The study population represents a typical geriatric oncologic cohort in a tertiary referral center.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2025-05-10 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
Postoperative Decision Satisfaction Score | From the day of surgery to postoperative day 15.
  Decision satisfaction will be assessed using the Decision Regret Scale (DRS) on postoperative day 15. The scale measures the patient's satisfaction with the surgical decision-making process, with higher scores indicating greater regret.

SECONDARY OUTCOMES:
Preoperative Cognitive Function (MoCA) | Up to 1 day before surgery
  Cognitive function will be evaluated preoperatively using the Montreal Cognitive Assessment (MoCA), which assesses multiple cognitive domains. Lower scores indicate worse cognitive performance.
Preoperative Physical Frailty (CFS) | Up to 1 day before surgery
  Physical frailty will be assessed preoperatively using the Clinical Frailty Scale (CFS), with higher scores indicating greater frailty.
Postoperative Adaptation Score | From the day of surgery to 30 days after surgery
  A composite adaptation score will be assessed to evaluate postoperative recovery and behavioral adaptation. This score includes parameters such as early postoperative mobilization (e.g., time to ambulation), respiratory exercises compliance (e.g., frequency of incentive spirometry use), medication adherence, attendance to scheduled follow-ups, and return to baseline functional status. Higher scores indicate better postoperative adaptation.
Length of Hospital Stay | From date of surgery until hospital discharge, assessed up to 14 days
  The number of days from the date of surgery to hospital discharge will be recorded as the length of hospital stay.
30-Day Postoperative Complications | Within 30 days after surgery
  Postoperative complications occurring within 30 days of surgery will be recorded and classified according to the Clavien-Dindo classification system.

CONTACTS AND LOCATIONS:
Overall Officials: Celal Akdemir, MD, Principal Investigator — Izmir City Hospital
Locations (1):
- İzmir City Hospital, Izmir, Turkey (Türkiye)